CLINICAL TRIAL: NCT00888524
Title: Evidence-Based Physiotherapy With and Without Deep Water Running on Non-Specific Low Back Pain. A Randomized Controlled Trial
Brief Title: Plus Deep Water Running on Low Back Pain
Acronym: +DWR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Jose Angel Narvaez Bueno, Vice_chancelor of Universoty of Malaga, research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 857 IAC 0630041300; 857 IAC 0630041300
Record Dates: First submitted 2009-04-22; First posted 2009-04-27 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Low Back Pain
Keywords: head out water immersion,; high intensity exercise,; evidence-based physiotherapy;; aquatics;; hydrotherapy; aquatics therapy; exercise therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General Practice (GP) in Physio plus Deep water running (Experimental): A supplementation of Deep Water running exercises of 20 minutes in high intensity around aerobic thresholds estimated in individual land and water test
  Interventions: Procedure: GP in Physio plus DWR
- General Practice in Physio (Experimental): A procedure of evidence-based physiotherapy is usual care in pragmatic trial
  Interventions: Procedure: GP in Physio

INTERVENTIONS:
Procedure: GP in Physio — manual therapy, educational advice of health promotion and physical exercises therapy based in a individual assessment
  Arms: General Practice in Physio
Procedure: GP in Physio plus DWR — GP in Physio plus a supplementation of DWR training in high intensive aerobic threshold
  Arms: General Practice (GP) in Physio plus Deep water running

SUMMARY:
Objectives: To evaluate the effect size on non-specific chronic low back pain (CLBP) of evidence-based physiotherapy (EBP) with and without the addition of deep water running (DWR) on pain, physical disability and general health state.

Materials and methods: Randomized, double-blind, controlled trial (therapists and assessors) involving 46 persons with CLBP over 15 weeks with two interventions, presented three times a week. Each group received EBP (personalized exercise program, manual therapy and health education) while one group performed supplementary 20 min sessions of DWR at the individualized aerobic threshold. Measurements were made pre and post intervention for pain, disability and general health. Range of motion of lumbar spine in the sagittal plane, maximum isometric strength and muscle endurance of lumbar and hip extensors was assessment.

ELIGIBILITY:
Inclusion Criteria:

* Participants were diagnosed with non-specific CLBP, with no radiation to the legs, and lasting at least three months

Exclusion Criteria:

* Low back pain as a result of specific spinal disease, infection, tumor, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome or caudal equine syndrome
* Patients not able to follow instructions
* Patients with any digressive condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
pain in VAS | scale 0 -100, pre and post intervention and follow up 6 and 12 month

SECONDARY OUTCOMES:
disability RMQ | scale 0-24, pre and post intervention and follow up 6 and 12 month
general (mental and physical) health state with SF-12 | scale 0 -100, pre and post intervention and follow up 6 and 12 month
functional Measurements: range on motion in degrees with inclinometer dual, strength with lineal dynamometer (newton) and endurance muscular with soerensen test (seconds) | scale physica of degrees, newtons and seconds pre post intervention and 6 and 12 month of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cuesta-Vargas, PhD, Principal Investigator — University of Malaga
Locations (1):
- School Medicine University of Malaga, Málaga, Malaga, Spain

REFERENCES:
- See also: University of Malaga — http://www.uma.es/
- See also: Research And Development of Spain — http://www.plannacionalidi.es/plan-idi-public/
- See also: Food and Drugs Administration — http://www.fda.gov/